CLINICAL TRIAL: NCT07282886
Title: Open-label, Prospective, Crossover, Proof-of-concept Study to Evaluate the Effect of Triple Therapy With Extrafine Beclomethasone Dipropionate/Formoterol Fumarate/Glycopyrrolate (BDP/FF/G) Via pMDI Compared With Non-extrafine Fluticasone Furoate/Umeclidinium/Vilanterol (FluF/UMEC/VI) Via DPI on Lung Ventilation and Clinical Outcomes in Subjects With Moderate to Severe Asthma
Brief Title: VENTURI (VENTilation Using Respiratory Imaging)
Acronym: VENTURI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Surya P Bhatt, MD, MSPH, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300015310; UAB (Other: UAB)
Record Dates: First submitted 2025-11-21; First posted 2025-12-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; fluticasone furoate; GSK573719; vilanterol

STUDY DESIGN:
Intervention Model Description: Single center, open-label, randomized crossover
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Randomized beclomethasone dipropionate/formoterol fumarate /glycopyrrolate (Experimental): For this randomized arm, Trimbow pMDI (BDP/FF/G 100/6/12.5 mcg), will be administered as two inhalations twice-daily 8 weeks following randomization.
  Interventions: Drug: Beclomethasone Dipropionate/Formoterol Fumarate/Glycopyrrolate pMDI
- Randomized fluticasone furoate/ umeclidinium/vilanterol (Active Comparator): For this randomized arm, Trelegy DPI (FluF/UMEC/VI 100/62.5/25 mcg), will be administered as one inhalation once daily for 8 weeks following randomization. .
  Interventions: Drug: Fluticasone Furoate/Umeclidinium/Vilanterol 100 MCG/1 ACTUATION-62.5 MCG/1 ACTUATION-25 MCG/1 ACTUATION Inhalation Powder
- Wash-Out (No Intervention): Following the 8-week treatment period, participants will be placed on an ICS/LABA therapy unrelated to study medications during a 4-week wash-out period prior to cross-over.
- Cross-Over beclomethasone dipropionate/formoterol fumarate /glycopyrrolate (Experimental): Following the washout period, participants that were randomized to receive Trelegy DPI (FluF/UMEC/VI 100/62.5/25 mcg) will be crossed over to receive Trimbow pMDI ( BDP/FF/G 100/6/12.5 mcg) for 8 weeks.
  Interventions: Drug: Beclomethasone Dipropionate/Formoterol Fumarate/Glycopyrrolate pMDI
- Cross-Over fluticasone furoate/ umeclidinium/vilanterol (Active Comparator): Following the washout period, participants that were randomized to receive Trimbow pMDI( BDP/FF/G 100/6/12.5 mcg) will be crossed over to receive Trelegy DPI (FluF/UMEC/VI 100/62.5/25 mcg) for 8 weeks.
  Interventions: Drug: Fluticasone Furoate/Umeclidinium/Vilanterol 100 MCG/1 ACTUATION-62.5 MCG/1 ACTUATION-25 MCG/1 ACTUATION Inhalation Powder

INTERVENTIONS:
Drug: Beclomethasone Dipropionate/Formoterol Fumarate/Glycopyrrolate pMDI — pMDI,100/6/12.5 mcg per inhalation
  Other Names: Trimbow; BDP/FF/G
  Arms: Cross-Over beclomethasone dipropionate/formoterol fumarate /glycopyrrolate; Randomized beclomethasone dipropionate/formoterol fumarate /glycopyrrolate
Drug: Fluticasone Furoate/Umeclidinium/Vilanterol 100 MCG/1 ACTUATION-62.5 MCG/1 ACTUATION-25 MCG/1 ACTUATION Inhalation Powder — Dry Powder Inhaler,100/62.5/25 mcg per inhalation
  Other Names: Trelegy Ellipta, 100 Mcg-62.5 Mcg-25 Mcg/Inh Inhalation Powder; FluF/UMEC/VI
  Arms: Cross-Over fluticasone furoate/ umeclidinium/vilanterol; Randomized fluticasone furoate/ umeclidinium/vilanterol

SUMMARY:
The purpose of the study is to enroll participants with uncontrolled asthma to evaluate the large and small airways and drug delivery utilizing two study drugs:

* Beclometasone dipropionate/Formoterol fumarate dihydrate/Glycopyrronium bromide (BDP/FF/G) or Trimbow
* Fluticasone furoate/Umeclidinium/Vilanterol (FluF/UMEC/VI ) or Trelegy Ellipta

DETAILED DESCRIPTION:
The study will comprise of 5 visits. A screening visit (V1, Week -2), with baseline assessment. At the randomization visit (V2, Week 0), patients will be randomized in a 1:1 ratio to receive one of the following treatments for 8 weeks:

* BDP/FF/G 100/6/12.5 mcg pMDI, two inhalations twice-daily
* FluF/UMEC/VI 100/62.5/25 mcg DPI, one inhalation once-daily

A subsequent visit will be performed at 8 weeks (V3), where participants will undergo spirometry, oscillometry, and imaging. Participants will then stop the assigned treatment and undergo a washout period of 4 weeks using an unrelated maintenance ICS/LABA combination inhaler.

Following the washout period, at the next visit (V4, Week 12) participants will then be crossed over to the other treatment they did not receive at randomization.

At the final visit (V5, Week 20), patients will once again undergo spirometry, oscillometry, and imaging. In the event of premature study discontinuation, an early termination (ET) visit will be conducted and the Investigator must fill in the "Study Termination" page in the eCRF, reporting the main reason for withdrawal.

Participants who were previously screened and found ineligible due to transient or correctable conditions (e.g., recent exacerbation) may be considered for rescreening twice. Rescreening must be approved by the Principal Investigator and documented in the subject's screening log.

Rescreening will follow the same procedures as the initial screening, including informed consent, unless otherwise specified in the protocol. The reason for rescreening and any changes in eligibility status must be clearly documented in the case report form (CRF) and source documents.

ELIGIBILITY:
Inclusion Criteria:

* Subject's written informed consent obtained prior to any study-related procedure.
* Patients aged ≥ 18 and ≤ 75 years
* Confirmed diagnosis of asthma (patients must have a documented history of asthma for at least 1 year with diagnosis before the age of 40 and/or pre-bronchodilator FEV1 between 50-80% of their predicted normal value, after appropriate washout from bronchodilators)
* Symptomatic on ICS/LABA treatment with ACT <20
* No exacerbations in the past 3 months requiring treatment with systemic corticosteroids or emergency department visit/ in-patient hospitalization
* The ability to be trained and correctly use a pressurized Meter Dose Inhaler (pMDI) and Dry Powder Inhaler (DPI)
* To have a cooperative attitude and the ability to perform the required outcomes measurements (e.g. spirometry maneuvers in sitting and supine position) and the ability to understand the risks involved
* WOCBP fulfilling one of the following criteria:

  1. WOCBP with fertile male partners: they and/or their partner must be willing to use a highly effective birth control method from the signature of the informed consent and until the follow-up visit or
  2. WOCBP with physician confirmed non-fertile male partners (contraception is not required in this case).
* Female patients of non-childbearing potential defined as physiologically incapable of becoming pregnant (i.e. post-menopausal or permanently sterile, e.g. amenorrheic for ≥12 consecutive months without alternative medical cause). Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. If indicated, as per investigator's request, post-menopausal status may be confirmed by follicle-stimulating hormone levels (according to local laboratory ranges).

Exclusion Criteria:

* Pregnant or lactating female
* Patients who had an exacerbation, defined as a sustained and acute deterioration of subject's symptoms and signs (dyspnea, cough and/or sputum production/purulence) that was either moderate, i.e. require treatment with systemic (oral/IV/IM) corticosteroids and/or antibiotics, or severe, i.e. require hospitalization, if their associated treatment/hospitalization occurred within 3 months prior to V1
* Inability to carry out pulmonary lung function testing, to comply with study procedures or with study treatment intake
* History of near fatal asthma or of a past hospitalization for asthma in intensive care unit which, in the judgement of the Investigator, may have placed the patient at undue risk
* Patients using systemic corticosteroid medication in the 4 weeks or slow-release corticosteroids in the 12 weeks, prior to screening
* Patients who suffer from COPD as defined by the current Global Initiative for Chronic Obstructive Lung Disease (GOLD) document
* History of a diagnosis of cystic fibrosis, bronchiectasis or alpha-1 antitrypsin deficiency, or any other significant lung disease which may have interfered with study evaluations
* Current smokers or current use of electronic cigarettes or ex-smokers with total cumulative exposure equal or more than 10 pack-years or having stopped smoking one year or less prior to screening visit
* Patients who had clinically significant cardiovascular condition according to investigator's judgement, such as but not limited to: congestive heart failure (NYHA class >2), acute ischemic heart disease in the last year prior to study screening, history of sustained cardiac arrhythmias or sustained and non-sustained cardiac arrhythmias diagnosed in the last 6 months (sustained meant lasting more than 30 seconds or ending only with external action, or led to hemodynamic collapse; non-sustained meant >3 beats <30 seconds, and or ending spontaneously, and or asymptomatic), high degree impulse conduction blocks (>2nd degree atrioventricular block type 2). Similarly, patients affected by persistent, long standing or paroxysmal AF were not considered for enrollment
* Patients who are unable to undergo imaging procedures for CT scans or MRI or demonstrate intolerance to Xenon gas
* Patients who have participated in a recent therapeutic trial (within past 6 months)
* Patients who have a milk protein allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of extrafine beclomethasone dipropionate/formoterol fumarate /glycopyrrolate compared with non-extrafine fluticasone furoate/ umeclidinium/vilanterol on ventilation defect percentage utilizing 129Xenon MRI. | 8 weeks
  Assess pre-post intervention ventilation defect percentage

SECONDARY OUTCOMES:
Investigating the association of small airways deposition on lung function | 8 weeks
  Test pre-post resistance on oscilometry and FEV1
Understanding the impact on asthma control using the Asthma Control Test | 8 Weeks
  Test pre-post change in Asthma Control Test

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States